CLINICAL TRIAL: NCT00071799
Title: A Multicenter, Randomized, Open-label, Parallel-group, Phase 3 Trial of Subcutaneous Azacitidine Plus Best Supportive Care Versus Conventional Care Regimens Plus Best Supportive Care for the Treatment of Myelodysplastic Syndromes (MDS)
Brief Title: A Survival Study in Patients With High Risk Myelodysplastic Syndromes Comparing Azacitidine Versus Conventional Care
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AZA PH GL 2003 CL001
Record Dates: First submitted 2003-10-31; First posted 2003-11-05 (Estimated); Results first posted 2010-07-05 (Estimated); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Azacitidine; Cytarabine; Anthracyclines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Azacitidine (Experimental): Study Drug plus best supportive care. Treatment with erythropoietin was not permitted
  Interventions: Drug: Azacitidine
- Conventional Care (Active Comparator): Physician choice of low dose cytarabine (plus best supportive care), standard chemotherapy (plus best supportive care) or best supportive care (only). Treatment with erythropoietin was not permitted
  Interventions: Other: Physician Choice

INTERVENTIONS:
Drug: Azacitidine — Azacitidine was injected subcutaneously (SC) at an initial dose of 75mg/m^2/day for 7 days. The 7-day dosing was repeated every 28 days with dose adjustment based on predefined hematology and renal laboratory results. Number of cycles: Azacitidine treatment was to be continued until the end of the study unless treatment was discontinued due to unacceptable toxicity, relapse after complete or partial response, transformation to AML or disease progression.
  Other Names: AZA
  Arms: Azacitidine
Other: Physician Choice — Physician Choice was one of three options:
  * Best supportive care (BSC) alone,
  * Low-dose cytarabine subcutaneously for 14 days every 28 to 42 days, or
  * Standard chemotherapy administered for induction as a continuous intravenous infusion of cytarabine over 7 days plus an anthracycline (daunorubicin, idarubicin, or mitoxantrone) on Days 1, 2, and 3; and, for those eligible, 1 or 2 consolidation cycles administered as continuous intravenous infusions of cytarabine for 3 to 7 days with the same anthracycline that was used at induction on Days 1 and 2 (each cycle between 28 to 70 days from the start of the previous cycle).
  All three options included best supportive care
  Other Names: cytarabine; anthracycline
  Arms: Conventional Care

SUMMARY:
The purpose of this study is to determine whether patients with high-risk myelodysplastic syndromes (MDS) treated with azacitidine have improved survival compared to conventional care treatments. The study will also assess the effect of treatments on response, duration of response, and transformation to acute myeloid leukemia (AML). The study will continue for 12 months following last patient enrolled.

See study AZA PH GL 2003 CL 001 E for information about the extension to this study.

DETAILED DESCRIPTION:
Comparison/Control Interventions offered the physician three options:

* Best supportive care (BSC) alone,
* Low-dose cytarabine subcutaneously for 14 days every 28 to 42 days, or
* Standard chemotherapy administered for induction as a continuous intravenous infusion of cytarabine over 7 days plus an anthracycline (daunorubicin, idarubicin, or mitoxantrone) on Days 1, 2, and 3; and, for those eligible, 1 or 2 consolidation cycles administered as continuous intravenous infusions of cytarabine for 3 to 7 days with the same anthracycline that was used at induction on Days 1 and 2 (each cycle between 28 to 70 days from the start of the previous cycle).

All three options included best supportive care. Neither the experimental group (azacitidine) nor any of the comparison/control options allowed use of erythropoietin.

Duration of Intervention: Patients will be treated until death, withdrawal, unacceptable toxicity or conclusion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of refractory anemia with excess blasts or refractory anemia with excess blasts in transformation according to the French-American-British classification system for myelodysplastic syndromes (MDS) and a relatively high risk of acute myeloid leukemia (AML) transformation, with an International Prognostic Scoring System score of INT-2 or High.
* Be 18 years of age or older
* Have a life expectancy of at least 3 months
* Be unlikely to proceed to bone marrow or stem cell transplantation therapy following remission
* Have serum bilirubin levels less than or equal to 1.5 times the upper limit of normal range for the laboratory
* Have serum glutamic-oxaloacetic transaminase (aspartate aminotransferase) or serum glutamic-pyruvic transaminase (alanine aminotransferase) levels less than or equal to 2 times the upper limit of normal (unless these are considered to be related to transfusion-induced secondary hemosiderosis)
* Have serum creatinine levels less than or equal to 1.5 times the upper limit of normal

Exclusion Criteria:

* Secondary myelodysplastic syndromes (MDS)
* Prior treatment with azacitidine;
* Prior history of acute myeloid leukemia (AML);
* Malignant disease diagnosed within prior 12 months;
* Metastatic disease;
* Hepatic tumors;
* Radiation, chemotherapy, cytotoxic therapy for non-MDS conditions within prior 12 months;
* Prior transplantation or cytotoxic therapy to treat MDS;
* Serious medical illness likely to limit survival to 12 months or less;
* Treatment with erythropoietin or myeloid growth factors during prior 21 days or androgenic hormones during prior 13 days;
* Active HIV, viral hepatitis type B or C;
* Treatment with investigational drugs during prior 30 days;
* Within the 28-day screening period, documented red cell folate deficiency, as evidenced by red blood cell folate (not serum folate) or vitamin B12 deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Actual)
Dates: Start 2003-11-01 (Actual); Primary Completion 2007-07-01 (Actual); Study Completion 2007-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: CL Beach, Study Director — Celgene Corporation
Locations (107):
- United States (8):
  - University of Alabama School of Medicine, Birmingham, Alabama
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Washington University School of Medicine, St Louis, Missouri
  - Mount Sinai Medical Center, New York, New York
  - Case Western Reserve University, Cleveland, Ohio
  - Oregon Cancer Center, Portland, Oregon
  - Western Pennsylvania Cancer Institute, Pittsburgh, Pennsylvania
  - Froedtert Memorial Lutheran Hospital, Milwaukee, Wisconsin
- Australia (10):
  - Liverpool Hospital, Liverpool, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - The Newcastle Mater Miseriecordiae Hospital, Warratah, New South Wales
  - Royal Brisbane Hospital, Hersten, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Peter MacCallum Cancer Institute, East Melbourne, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - The Royal Perth Hospital, Perth, Western Australia
- Bulgaria (6):
  - First Clinical Base - Clinic of Hematology, MHAT - Pleven, Pleven
  - MHAT "St George" Clinic of Hematology, Plovdiv, Plovdiv
  - III-rd Internal Department, District Dispensary for Oncology diseases with stationary(DDOncDIU), Plovdiv
  - National Centre of Hematology and Transfusiology, Sofia, Sofia
  - Multiprofile Hospital for Active Treatment (MHAT), "St. Marina" Clinic of Hematology, Varna
  - University Multiprofile Hospital for Active Treatment "Sveta Marina", Varna
- Czechia (5):
  - Fakultni nemocnice Brno, Jihlavska, Brno
  - Fakultni nemocnice Hradec Kralove, Sokolska, Hradec Kralove
  - Fakultni Nemocnice Olomouc, Olomouc
  - Vseobecna Fakultni Nemocnice, Prague
  - Uslav Hematologie a Krevni Transfuze, Prague
- France (10):
  - Chu D'Angers, Angers
  - Hopital Beaujon, Clichy
  - Che De Lille, Lille
  - Hospital Edouard Herriot, Lyon
  - Institute Paoli Calmettes, Marseille
  - Chu De Nantes, Nantes
  - Hospital Saint Louis, Paris
  - Hopital Cochin, Paris
  - Centre Henri Becquerel, Rouen
  - Chu Purpan, Toulouse
- Germany (12):
  - Universitatsklinikum Benjamin Franklin, Hindenburgdamm, State of Berlin
  - Universitatsklinikum Bonn, Bonn
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Universitatsklinikum Carl Gustav Carus, Dresden
  - St Johannes Hospital, Duisburg
  - Heinrich-Heine University Dusseldorf, Düsseldorf
  - University Essen, Essen
  - Gerorg-August-Universitat Gottingen, Göttingen
  - Allgemeines Krankenhaus St. Georg, Hamburg
  - Universitatsklinikum Hambur-Eppendorf, Hamburg
  - Universitatsklinikum Kiel II, Kiel
  - Universitatsklinikum Ulm, Ulm
- Greece (6):
  - University Hospital-Attikon, Haidari, Athens
  - University General Hospital of Heraklio Voutes, Heraklio, Crete
  - District General Hospital of Athens, Athens
  - General Hospital of Chest Disease, Athens
  - University General Hospital of Ioannina, Ioannina
  - University General Hospital of Patra Rio, Pátrai
- Hungary (3):
  - Orszagos Gyogyintezeti Kozpont, Budapest
  - University of Pecs, 1st Dept of Internal Medicine, Pécs
  - University of Szeged, 2nd Department of Internal Medicine, Szeged
- Italy (10):
  - Policlinico S. Orsola-Malpighi, Bologna
  - Universita di Firenze, Florence
  - Ospedale San Martino, Genova
  - Instituto Nazionale Dei Tumori, Milan
  - Centro Oncologico Modenese, Modena
  - Ospedale San Eugenio, Roma
  - Policlinico Gemelli, Roma
  - Instituto Nazionale Tumori "Regina Elena", Roma
  - Ospedale Casa Sollievo Della Sofferenza - Irrc, San Giovanni Rotondo
  - Universita Degli Studi Di Sassari, Sassari
- Netherlands (2):
  - VU University Medical Center Amsterdam, Amsterdam
  - Univ Hospital St. Radboud, Nijmejen
- Poland (6):
  - Samodzielny Publiczny Szpital Kliniczny Nr 1, Gdansk
  - Wojewodzki Szpital Specjalistyczny, Lodz
  - Samodzielny Publiczny Szpital Kliniczny, Lublin
  - Wojskowy Instytut Medyczny, Warsaw
  - Samodzelny Publiczny Centralny Szpital Kliniczny, Warsaw
  - Samodzielny Publiczny Szpital Kliniczny Nr 1, Wroclaw
- Russia (6):
  - Burdenko Central Military Clinical Hospital, Moscow
  - Blokhin Cancer Research Center, Moscow
  - Scientific Haematology Center, Moscow, Moscow
  - Institute of Haematology & Blood Transfusion, Saint Petersburg
  - Pavlov State Medical University, Saint Petersburg
  - City Hospital #31, Saint Petersburg
- Spain (11):
  - Hospital Santa Creu I Sant Pau, Barcelona
  - Hospital Clinic, Barcelona
  - Hospital Universitario Germans Trias I Pujol, Barcelona
  - Hospital de Leon, León
  - Hospital Universitario De La Princesa, Madrid
  - Hospital Ramon Y Cajal, Madrid
  - Hospital La Paz, Madrid, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Son Llatzer, Palma de Mallorca
  - Hospital Universitario Del Salamanca, Salamanca
  - Hospital Universitario La Fe, Valencia
- Sweden (5):
  - Sahlgrenska University Hospital, Gothenburg
  - Lund Universtiy Hospital, Lund
  - University Hospital MAS, Malmo
  - Huddinge University Hospital, Stockholm
  - Uppsala University Hospital, Uppsala
- United Kingdom (7):
  - Royal Bournemouth General Hospital, Bournemouth
  - St. Bartholomew's Hospital, London
  - Kings College Hospital NHS Trust, London
  - Christie Hospital, Manchester
  - Norfolk and Norwich University Hospital, Norwich
  - John Radcliffe Hospital, Oxford
  - Royal Cornwall Hospital, Truro

REFERENCES:
- [Result] Fenaux P, Mufti GJ, Hellstrom-Lindberg E, Santini V, Gattermann N, Germing U, Sanz G, List AF, Gore S, Seymour JF, Dombret H, Backstrom J, Zimmerman L, McKenzie D, Beach CL, Silverman LR. Azacitidine prolongs overall survival compared with conventional care regimens in elderly patients with low bone marrow blast count acute myeloid leukemia. J Clin Oncol. 2010 Feb 1;28(4):562-9. doi: 10.1200/JCO.2009.23.8329. Epub 2009 Dec 21. PMID 20026804
- [Result] Fenaux P, Gattermann N, Seymour JF, Hellstrom-Lindberg E, Mufti GJ, Duehrsen U, Gore SD, Ramos F, Beyne-Rauzy O, List A, McKenzie D, Backstrom J, Beach CL. Prolonged survival with improved tolerability in higher-risk myelodysplastic syndromes: azacitidine compared with low dose ara-C. Br J Haematol. 2010 Apr;149(2):244-9. doi: 10.1111/j.1365-2141.2010.08082.x. Epub 2010 Feb 5. PMID 20136825
- [Result] Santini V, Fenaux P, Mufti GJ, Hellstrom-Lindberg E, Silverman LR, List A, Gore SD, Seymour JF, Backstrom J, Beach CL. Management and supportive care measures for adverse events in patients with myelodysplastic syndromes treated with azacitidine*. Eur J Haematol. 2010 Aug;85(2):130-8. doi: 10.1111/j.1600-0609.2010.01456.x. Epub 2010 Apr 12. PMID 20394651
- [Result] Seymour JF, Fenaux P, Silverman LR, Mufti GJ, Hellstrom-Lindberg E, Santini V, List AF, Gore SD, Backstrom J, McKenzie D, Beach CL. Effects of azacitidine compared with conventional care regimens in elderly (>/= 75 years) patients with higher-risk myelodysplastic syndromes. Crit Rev Oncol Hematol. 2010 Dec;76(3):218-27. doi: 10.1016/j.critrevonc.2010.04.005. Epub 2010 May 6. PMID 20451404
- [Result] Fenaux P, Mufti GJ, Hellstrom-Lindberg E, Santini V, Finelli C, Giagounidis A, Schoch R, Gattermann N, Sanz G, List A, Gore SD, Seymour JF, Bennett JM, Byrd J, Backstrom J, Zimmerman L, McKenzie D, Beach C, Silverman LR; International Vidaza High-Risk MDS Survival Study Group. Efficacy of azacitidine compared with that of conventional care regimens in the treatment of higher-risk myelodysplastic syndromes: a randomised, open-label, phase III study. Lancet Oncol. 2009 Mar;10(3):223-32. doi: 10.1016/S1470-2045(09)70003-8. Epub 2009 Feb 21. PMID 19230772
- [Derived] Gore SD, Fenaux P, Santini V, Bennett JM, Silverman LR, Seymour JF, Hellstrom-Lindberg E, Swern AS, Beach CL, List AF. A multivariate analysis of the relationship between response and survival among patients with higher-risk myelodysplastic syndromes treated within azacitidine or conventional care regimens in the randomized AZA-001 trial. Haematologica. 2013 Jul;98(7):1067-72. doi: 10.3324/haematol.2012.074831. Epub 2013 Apr 12. PMID 23585522
- See also: Study record for the extension study of AZA PH GL 2003 CL 001 — http://www.clinicaltrials.gov/ct2/show/NCT01186939?term=NCT01186939&rank=1

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 738 patients screened from 98 investigator sites. Randomized patients contributed by 79 investigator sites.
Groups:
- Azacitidine: Azacitidine, 75 mg/m^2/day given by subcutaneous injection for 7 days of every 28 day cycle, plus best supportive care.
- Conventional Care: Physician choice of low dose cytarabine, standard chemotherapy, or best supportive care (consisting of blood products, growth factors, antibiotics)
Period: Overall Study
Arm/Group | Azacitidine | Conventional Care
Started | 179 | 179 (Best supportive care: 105, Low-dose cytarabine: 49, Standard chemotherapy: 25 patients)
Completed | 109 (Includes those who died or transformed to AML, or receiving drug + eligible for extension period.) | 81 (Includes patients who died or transformed to AML during treatment, or were still receiving drug.)
Not Completed | 70 | 98
Not completed — Adverse Event | 19 | 10
Not completed — Protocol Violation | 1 | 7
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 15 | 37
Not completed — Physician Decision | 0 | 2
Not completed — Lack of Efficacy | 11 | 18
Not completed — Disease Progression | 23 | 20
Not completed — Different Central+Local Pathology Review | 0 | 1
Not completed — Not Documented | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azacitidine | Conventional Care | Total
Number analyzed (Participants) | 179 | 179 | 358
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.0 (7.57) | 69.2 (7.87) | 68.6 (7.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 60 | 107
  Male | 132 | 119 | 251
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 177 | 175 | 352
  Black or African American | 0 | 0 | 0
  Asian/Oriental | 2 | 3 | 5
  Hispanic | 0 | 1 | 1
  Other | 0 | 0 | 0
French-American-British (FAB) Classification [Number; unit: participants] — FAB classifications were determined by the Independent Review Committee
  participants
    Refractory anemia with excess blasts (RAEB) | 104 | 103 | 207
    RAEB in transformation | 61 | 62 | 123
    Modified chronic myelomonocytic leukemia | 6 | 5 | 11
    Acute myeloid leukemia | 1 | 1 | 2
    Myeloproliferative disease | 4 | 2 | 6
    Indeterminate | 3 | 6 | 9
International Prognostic Scoring System (IPSS) [Number; unit: participants] — The international prognostic scoring system (IPSS) is a standard for risk assessment in primary myelodysplastic syndromes (MDS) that categorizes prognoses taking into account cytogenetics, cytopenias, blasts and blood counts. The scale is 0-3.5 at .5 increments. Scores of 2.5-3.5 represent high risk which corresponds to poorer prognosis. The assessment was performed by the Independent Review Committee.
  participants
    Intermediate risk level 1 (0.5-1.0) | 5 | 13 | 18
    Intermediate risk level 2 (1.5-2.0) | 76 | 70 | 146
    High risk (2.5-3.5) | 82 | 85 | 167
    Not applicable | 5 | 3 | 8
    Indeterminate | 11 | 8 | 19
World Health Organization (WHO) Classification [Number; unit: participants] — WHO classifications were determined by the Independent Review Committee
  participants
    Refractory anemia with excess blasts - 1 | 14 | 17 | 31
    Refractory anemia with excess blasts - 2 | 98 | 95 | 193
    Chronic myelomonocytic leukemia - 1 (CMMoL-1) | 1 | 0 | 1
    Chronic myelomonocytic leukemia - 2 (CMMoL-2) | 10 | 5 | 15
    Acute myeloid leukemia | 55 | 58 | 113
    Indeterminate | 1 | 4 | 5
Body Surface Area [Mean (Standard Deviation); unit: meters squared] | 1.9 (0.19) | 1.8 (0.19) | 1.9 (0.19)
Weight [Mean (Standard Deviation); unit: kilograms] | 76.5 (14.08) | 74.6 (13.58) | 75.6 (13.85)

OUTCOME MEASURES:

1. Primary Outcome: Kaplan-Meier Estimates for Median Time to Death From Any Cause
Description: Kaplan-Meier estimates for the median months until death from any cause within the intent-to-treat population. Patients surviving at the end of the follow-up period were censored at the date of last contact. If a patient withdrew consent to follow-up or was lost to follow-up, the patient was censored as of the last date of contact.
Time Frame: Day 1 (randomization) to 42 months
Population: Intent to treat population. Includes participants who died and participants who were censored.
Measure: Number; unit: months
Arm/Group | Azacitidine | Conventional Care
Number analyzed (Participants) | 179 | 179
months | 24.46 | 15.02
Statistical Analysis 1: Comparison: Azacitidine vs Conventional Care; A 95% CI range value of 'does not exist' is not accommodated in the results table, so all the 95% CI range values are offered here. Azacitidine: low range of 17.9 months and high range of 'does not exist'. Conventional Care: low range of 9.8 and high range of 17.0 months; Test type: Superiority or Other; p = 0.0001, Log Rank; The p value is two-sided from the log rank test stratified by the randomization stratification factors of IPSS classification and FAB classification
Statistical Analysis 2: Comparison: Azacitidine vs Conventional Care; Test type: Superiority or Other; p = 0.0002, Regression, Cox; Hazard Ratio (HR) = 0.58, 95% CI 2-sided [0.43 to 0.77] — Cox proportional hazards model stratified on the randomization factors of FAB and IPSS with model term of treatment

2. Primary Outcome: Summary of Subgroup Analyses for Kaplan-Meier Estimates for Time to Death From Any Cause
Description: Kaplan-Meier estimates for the median months until death from any cause within the intent-to-treat population. Patients surviving at the end of the follow-up period were censored at the date of last contact. If a patient withdrew consent to follow-up or was lost to follow-up, the patient was censored as of the last date of contact.
  Subgroups that were analyzed are age, gender, French-American-British (FAB) classification, World Health Organization (WHO) classification and International Prognostic Scoring System (IPSS) classification.
Time Frame: Day 1 (randomization) to 42 months
Population: Intent to treat population. Includes participants who died and those who were censored.
Measure: Number; unit: months
Arm/Group | Azacitidine | Conventional Care
Number analyzed (Participants) | 179 | 179
months
  Age <65 years | 11.31 | 7.87
  Age >= 65 years | 24.46 | 13.87
  Age >= 75 years | 8.92 | 6.20
  Gender: Male | 24.46 | 15.02
  Gender: Female | 25.11 | 14.85
  FAB: Refractory anemia with excess blasts (RAEB) | 34.66 | 15.21
  FAB: RAEB in transformation | 17.25 | 15.25
  WHO: RAEB 1 | 11.54 | 6.72
  WHO: RAEB 2 | 21.11 | 15.02
  WHO: Other (AML, CMMoL-1 and 2, indeterminate) | 20.46 | 15.25
  IPSS: Intermediate 2 | 34.66 | 16.89
  IPSS: High | 19.21 | 14.52
Statistical Analysis 1: Comparison: Azacitidine vs Conventional Care; Age < 65 years The Kaplan-Meier median time to death was not reached due to a small number of events, so the KM 25th percentile survival time is presented. Some of the values in outcome table #2 do not have 95% CI values so no 95% CI ranges are contained in the table. Those 95% CI ranges are added here. Azacitidine: low range of 7.1 months and high range of 15.6 months. Conventional Care: low range of 4.4 and high range of 12.4 months; Test type: Superiority or Other; p = 0.3973, Log Rank — The p value is two-sided from the log rank test stratified by the randomization stratification factors of IPSS classification and FAB classification
Statistical Analysis 2: Comparison: Azacitidine vs Conventional Care; Age >= 65 years Some of the values in outcome table #2 do not have 95% CI values so no 95% CI ranges are contained in the table. Those 95% CI ranges are added here. Azacitidine: low range of 17.1 months and high range of 34.7 months. Conventional Care: low range of 8.8 and high range of 16.4 months; Test type: Superiority or Other; p < 0.0001, Log Rank — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Azacitidine vs Conventional Care; Age >= 75 years. The Kaplan-Meier median time to death was not reached due to a small number of events, so the KM 25th percentile survival time is presented. Some of the values in outcome table #2 do not have 95% CI values so no 95% CI ranges are contained in the table. Those 95% CI ranges are added here. Azacitidine: low range of 1.7 months and high range of 15.0 months. Conventional Care: low range of 4.1 and high range of 7.6 months; Test type: Superiority or Other; p = 0.0707, Log Rank — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Azacitidine vs Conventional Care; Gender: Male Some of the values in outcome table #2 do not have 95% CI values so no 95% CI ranges are contained in the table. Those 95% CI ranges are added here. Azacitidine: low range of 17.9 months and high range of 'does not exist'. Conventional Care: low range of 10.8 and high range of 17.2 months; Test type: Superiority or Other; p = 0.0042, Log Rank — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Azacitidine vs Conventional Care; Gender: Female Some of the values in outcome table #2 do not have 95% CI values so no 95% CI ranges are contained in the table. Those 95% CI ranges are added here. Azacitidine: low range of 13.0 months and high range of 'does not exist'. Conventional Care: low range of 8.2 and high range of 17.6 months; Test type: Superiority or Other; p = 0.0469, Log Rank — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: Azacitidine vs Conventional Care; FAB: Refractory anemia with excess blasts (RAEB). All patients were stratified at randomization by FAB classification and IPSS score as determined by the investigator using centrally read bone marrow and cytogenetic data. Subsequently, the FAB classifications and IPSS scores were reviewed by an Independent Review Committee (IRC). The subgroup analyses presented by FAB and IPSS represent the FAB classification and IPSS scores as determined by the IRC; Test type: Superiority or Other; p = 0.0056, Log Rank — 95% CI ranges are added here. Azacitidine: low range of 21.1 months and high range of 'does not exist'. Conventional Care: low range of 9.3 and high range of 21.9 months; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Azacitidine vs Conventional Care; FAB: RAEB in transformation Some of the values in outcome table #2 do not have 95% CI values so no 95% CI ranges are contained in the table. Those 95% CI ranges are added here. Azacitidine: low range of 11.7 months and high range of 'does not exist'. Conventional Care: low range of 9.4 and high range of 17.0 months; Test type: Superiority or Other; p = 0.0322, Log Rank — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 8: Comparison: Azacitidine vs Conventional Care; WHO: RAEB 1. The Kaplan-Meier median time to death was not reached due to a small number of events, so the KM 25th percentile survival time is presented. Some of the values in outcome table #2 do not have 95% CI values so no 95% CI ranges are contained in the table. Those 95% CI ranges are added here. Azacitidine: low range of 6.6 months and high range of 'does not exist'. Conventional Care: low range of 1.8 and high range of 9.8 months; Test type: Superiority or Other; p = 0.1679, Log Rank — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 9: Comparison: Azacitidine vs Conventional Care; WHO: RAEB-2 Some of the values in outcome table #2 do not have 95% CI values so no 95% CI ranges are contained in the table. Those 95% CI ranges are added here. Azacitidine: low range of 15.9 months and high range of 'does not exist'. Conventional Care: low range of 8.8 and high range of 19.4 months; Test type: Superiority or Other; p = 0.0692, Log Rank — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 10: Comparison: Azacitidine vs Conventional Care; WHO: Other Some of the values in outcome table #2 do not have 95% CI values so no 95% CI ranges are contained in the table. Those 95% CI ranges are added here. Azacitidine: low range of 15.6 months and high range of 'does not exist'. Conventional Care: low range of 11.1 and high range of 17.5 months; Test type: Superiority or Other; p = 0.0017, Log Rank — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 11: Comparison: Azacitidine vs Conventional Care; IPSS: Intermediate 2 All patients were stratified at randomization by FAB classification and IPSS score as determined by the investigator using centrally read bone marrow and cytogenetic data. Subsequently, the FAB classifications and IPSS scores were reviewed by an Independent Review Committee (IRC). The subgroup analyses presented by FAB and IPSS represent the FAB classification and IPSS scores as determined by the IRC; Test type: Superiority or Other; p = 0.1030, Log Rank — 95% CI ranges are added here. Azacitidine: low range of 17.1 months and high range of 'does not exist'. Conventional Care: low range of 8.7 and high range of 24.1 months; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: Azacitidine vs Conventional Care; IPSS: High All patients were stratified at randomization by FAB classification and IPSS score as determined by the investigator using centrally read bone marrow and cytogenetic data. Subsequently, the FAB classifications and IPSS scores were reviewed by an Independent Review Committee (IRC). The subgroup analyses presented by FAB and IPSS represent the FAB classification and IPSS scores as determined by the IRC; Test type: Superiority or Other; p = 0.0020, Log Rank — 95% CI ranges are added here. Azacitidine: low range of 15.0 months and high range of 'does not exist'. Conventional Care: low range of 9.0 and high range of 17.0 months; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Kaplan-Meier Estimate for Median Time to Transformation to Acute Myeloid Leukemia (AML) or Death From Any Cause, Whichever Occurred First
Description: The time to transformation to AML or death from any cause (whichever occurred first) was defined as the number of days from the date of randomization until the date of documented AML transformation or death from any cause. Patients who did not transform to AML or die were censored at the date of last follow-up.
Time Frame: Day 1 (randomization) to 42 months
Population: Intent to treat population. Participants who either transformed to AML or died are 120 for azacitidine and 132 for conventional care. Remaining participants were censored.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Azacitidine | Conventional Care
Number analyzed (Participants) | 179 | 179
months | 13.02 [9.9 to 15.0] | 7.61 [5.4 to 9.8]
Statistical Analysis 1: Comparison: Azacitidine vs Conventional Care; Test type: Superiority or Other; p = 0.0025, Log Rank — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Azacitidine vs Conventional Care; Test type: Superiority or Other; p = 0.0027, Regression, Cox; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.53 to 0.87] — Cox proportional hazards model stratified on the randomization factors of FAB and IPSS with model term of treatment

4. Secondary Outcome: Kaplan-Meier Estimates for Median Time to Transformation to Acute Myeloid Leukemia (AML)
Description: The time to transformation to AML was defined as the number of days from the date of randomization until the date of documented AML transformation, defined as a bone marrow blast count ≥ 30% independent of baseline bone marrow count. Patients who did not transform to AML were censored at the date of last follow-up or date of death.
Time Frame: Day 1 (randomization) to 42 months
Population: Intent to treat population. Participants who were transformed to AML are 78 for azacitidine and 71 for conventional care. Remaining participants were censored based on the last bone marrow assessment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Azacitidine | Conventional Care
Number analyzed (Participants) | 179 | 179
months | 20.66 [14.9 to 25.5] | 15.44 [12.4 to 22.5]
Statistical Analysis 1: Comparison: Azacitidine vs Conventional Care; Test type: Superiority or Other; p = 0.2555, Log Rank — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Azacitidine vs Conventional Care; Test type: Superiority or Other; p = 0.2562, Regression, Cox; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.60 to 1.15] — Cox proportional hazards model stratified on the randomization factors of FAB and IPSS with model term of treatment

5. Secondary Outcome: Summary of Participants' Red Blood Cell (RBC) Transfusion Status for Participants Who Were Transfusion Dependent at Baseline
Description: Summary of dependence and independence from red blood cell (RBC) transfusion at baseline and during treatment, for patients who were dependent at baseline. A patient was considered transfusion independent at baseline if the patient had no transfusions during the 56 days prior to randomization. During study, a patient was considered transfusion independent during the on-treatment period if the patient had no transfusions during any 56 consecutive days or more. Otherwise, the patient was considered transfusion dependent.
Time Frame: Day 1 (randomization) to 42 months
Population: Intent to treat population
Measure: Number; unit: participants
Arm/Group | Azacitidine | Conventional Care
Number analyzed (Participants) | 111 | 114
participants
  Baseline Dependent; On-Treatment Independent | 50 | 13
  Baseline Dependent; On-Treatment Dependent | 61 | 101
Statistical Analysis 1: Comparison: Azacitidine vs Conventional Care; The p value is from Fisher's exact test comparing the difference in the azacitidine group and the combined group of CCR regimens among patients who were transfusion dependent at baseline and transfusion independent during the on-treatment period; Test type: Superiority or Other; p < 0.0001, Fisher Exact

6. Secondary Outcome: Summary of Participants' Red Blood Cell (RBC) Transfusion Status for Participants Who Were Transfusion Independent at Baseline
Description: Summary of dependence and independence from red blood cell (RBC) transfusion at baseline and during treatment, for patients who were independent at baseline. A patient was considered transfusion independent at baseline if the patient had no transfusions during the 56 days prior to randomization. During study, a patient was considered transfusion independent during the on-treatment period if the patient had no transfusions during any 56 consecutive days or more. Otherwise, the patient was considered transfusion dependent.
Time Frame: Day 1 (randomization) to 42 months
Population: Intent to treat population
Measure: Number; unit: participants
Arm/Group | Azacitidine | Conventional Care
Number analyzed (Participants) | 68 | 65
participants
  Baseline Independent; On-Treatment Independent | 58 | 37
  Baseline Independent; On-Treatment Dependent | 10 | 28
Statistical Analysis 1: Comparison: Azacitidine vs Conventional Care; The p value is from Fisher's exact test comparing the difference in the azacitidine group and the combined group of CCR regimens among patients who were transfusion independent at baseline and remained transfusion independent during the on-treatment period; Test type: Superiority or Other; p = 0.0005, Fisher Exact

7. Secondary Outcome: Summary of Participants' Platelet Transfusion Status for Participants Who Were Transfusion Dependent at Baseline
Description: Summary of dependence and independence from platelet transfusion at baseline and during treatment for patients who were dependent at baseline. A patient was considered transfusion independent at baseline if the patient had no transfusions during the 56 days prior to randomization. During study, a patient was considered transfusion independent during the on-treatment period if the patient had no transfusions during any 56 consecutive days or more. Otherwise, the patient was considered transfusion dependent.
Time Frame: Day 1 (randomization) to 42 months
Population: Intent to treat population
Measure: Number; unit: participants
Arm/Group | Azacitidine | Conventional Care
Number analyzed (Participants) | 38 | 27
participants
  Baseline Dependent; On-Treatment Independent | 16 | 11
  Baseline Dependent; On-Treatment Dependent | 22 | 16
Statistical Analysis 1: Comparison: Azacitidine vs Conventional Care; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 1.000, Fisher Exact

8. Secondary Outcome: Summary of Participants' Platelet Transfusion Status for Participants Who Were Transfusion Independent at Baseline
Description: Summary of dependence and independence from platelet transfusion at baseline and during treatment for patients who were independent at baseline. A patient was considered transfusion independent at baseline if the patient had no transfusions during the 56 days prior to randomization. During study, a patient was considered transfusion independent during the on-treatment period if the patient had no transfusions during any 56 consecutive days or more. Otherwise, the patient was considered transfusion dependent.
Time Frame: Day 1 (randomization) to 42 months
Population: Intent to treat population
Measure: Number; unit: participants
Arm/Group | Azacitidine | Conventional Care
Number analyzed (Participants) | 141 | 152
participants
  Baseline Independent; On-Treatment Independent | 126 | 102
  Baseline Independent; On-Treatment Dependent | 15 | 50
Statistical Analysis 1: Comparison: Azacitidine vs Conventional Care; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p < 0.0001, Fisher Exact

9. Secondary Outcome: Number of Participants Considered Hematologic Responders by Investigator Determinations Using International Working Group (IWG 2000) Criteria for Myelodysplastic Syndrome (MDS)
Description: Investigator determined responses followed IWG criteria for
  * complete remission(CR): repeat bone marrow show <5% myeloblasts, and peripheral blood evaluations lasting >=2 months of hemoglobin(>110 g/L), neutrophils(>=1.5x10^9/L), platelets(>=100x10^9/L), blasts (0%) and no dysplasia
  * partial remission(PR) is the same as CR for peripheral blood: bone marrow shows blasts decrease by >=50% or a less advanced FAB classification from pretreatment
  * stable disease(SD) is a failure to achieve at least a partial remission, but with no evidence of progression for at least 2 months.
Time Frame: Day 1 to 42 months
Population: Intent to treat population.
Measure: Number; unit: participants
Arm/Group | Azacitidine | Conventional Care
Number analyzed (Participants) | 179 | 179
participants
  Overall (Complete + Partial Remission) | 51 | 21
  Complete Remission | 30 | 14
  Partial Remission | 21 | 7
  Stable Disease | 75 | 65
Statistical Analysis 1: Comparison: Azacitidine vs Conventional Care; Overall (Complete + Partial Remission); Test type: Superiority or Other; p = 0.0001, Fisher Exact
Statistical Analysis 2: Comparison: Azacitidine vs Conventional Care; Complete remission; Test type: Superiority or Other; p = 0.0150, Fisher Exact
Statistical Analysis 3: Comparison: Azacitidine vs Conventional Care; Partial Remission; Test type: Superiority or Other; p = 0.0094, Fisher Exact
Statistical Analysis 4: Comparison: Azacitidine vs Conventional Care; Stable Disease; Test type: Superiority or Other; p = 0.3297, Fisher Exact

10. Secondary Outcome: Number of Participants Showing Hematologic Improvement Using International Working Group (IWG 2000) Criteria for Myelodysplastic Syndrome (MDS) Assessed by Independent Review Committee
Description: IWG 2000 Criteria: Pretreatment=hemoglobin <100g/L or RBC transfusion-dependent, platelet count <100x10^9/L or platelet transfusion dependent, absolute neutrophil count <1.5x10^9/L.
  Erythroid response: Major->20g/L increase or transfusion independent. Minor- 10-20g/L increase or >=50% decrease in transfusion requirements.
  Platelet response: Major-absolute increase of >=30x10^9/L or platelet transfusion independence. Minor->=50% increase.
  Neutrophil response: Major->=100% increase or an absolute increase of >0.5x10^9/L. Minor->=100% increase and absolute increase of <0.5x10^9/L.
Time Frame: Day 1 to 42 months
Population: Intent to treat population.
Measure: Number; unit: participants
Arm/Group | Azacitidine | Conventional Care
Number analyzed (Participants) | 179 | 179
participants
  Any Improvement n=177, 178 | 87 | 51
  Erythroid Response - Major n=157, 160 | 62 | 17
  Erythroid Response - Minor n=157, 160 | 2 | 1
  Platelet Response - Major n=141, 129 | 46 | 18
  Platelet Response - Minor n=138, 127 | 6 | 4
  Neutrophil Response - Major n=131, 111 | 25 | 20
  Neutrophil Response - Minor n=131, 111 | 5 | 9
Statistical Analysis 1: Comparison: Azacitidine vs Conventional Care; Any Improvement; Test type: Superiority or Other; p < 0.0001, Fisher Exact
Statistical Analysis 2: Comparison: Azacitidine vs Conventional Care; Erythroid Response - Major; Test type: Superiority or Other; p < 0.0001, Fisher Exact
Statistical Analysis 3: Comparison: Azacitidine vs Conventional Care; Erythroid Response - Minor; Test type: Superiority or Other; p = 0.6203, Fisher Exact
Statistical Analysis 4: Comparison: Azacitidine vs Conventional Care; Platelet Response - Major; Test type: Superiority or Other; p = 0.0003, Fisher Exact
Statistical Analysis 5: Comparison: Azacitidine vs Conventional Care; Platelet Response - Minor; Test type: Superiority or Other; p = 0.7514, Fisher Exact
Statistical Analysis 6: Comparison: Azacitidine vs Conventional Care; Neutrophil Response - Major; Test type: Superiority or Other; p = 0.8695, Fisher Exact
Statistical Analysis 7: Comparison: Azacitidine vs Conventional Care; Neutrophil Response - Minor; Test type: Superiority or Other; p = 0.1760, Fisher Exact

11. Secondary Outcome: Time to Disease Progression, Relapse After Complete or Partial Remission, or Death From Any Cause
Description: The time to disease progression, relapse after complete or partial remission (CR, PR), or death from any cause was defined as the time from the date of randomization until the first date of documented disease progression, relapse after CR or PR, or death from any cause.
Time Frame: Day 1 (randomization) to 42 months
Population: Intent to treat population. The number of participants with disease progression, relapse after remission or death from any cause is 84 for azacitidine and 79 for conventional care. Remaining participants were censored.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Azacitidine | Conventional Care
Number analyzed (Participants) | 179 | 179
months | 14.13 [9.5 to 27.6] | 8.82 [6.4 to 12.4]
Statistical Analysis 1: Comparison: Azacitidine vs Conventional Care; Test type: Superiority or Other; p = 0.0466, Log Rank — The p value is two-sided from the log rank test which compares whether the azacitidine and control group follow the same duration curve
Statistical Analysis 2: Comparison: Azacitidine vs Conventional Care; Test type: Superiority or Other; p = 0.0474, Regression, Cox; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.53 to 1.00]

12. Secondary Outcome: Duration of Any Hematologic Improvement
Description: The duration of improvement was defined as the time from the date of hematologic improvement until the date of first documented progression or relapse after hematologic improvement or death from any cause.
Time Frame: Day 1 (randomization) to 42 months
Population: Intent to treat population. Participants showing hematologic improvement were 48 in azacitidine and 31 in conventional care.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Azacitidine | Conventional Care
Number analyzed (Participants) | 87 | 51
months | 13.57 [10.1 to 16.3] | 5.18 [4.1 to 9.7]
Statistical Analysis 1: Comparison: Azacitidine vs Conventional Care; Test type: Superiority or Other; p = 0.0002, Log Rank — [p-value comment as in outcome 11, analysis 1]

13. Secondary Outcome: Number of Infections Per Treatment Year Requiring Intravenous Antibiotics, Antifungals or Antivirals
Description: The on-treatment adverse event rate of infection requiring IV antibiotics, antifungals, or antivirals per patient-years. The on-treatment period was considered the period from the date of randomization to the last treatment study visit.
Time Frame: Day 1 (randomization) to 42 months
Population: Intent to treat population
Measure: Number; unit: infections per treatment year
Arm/Group | Azacitidine | Conventional Care
Number analyzed (Participants) | 179 | 179
infections per treatment year | 0.16 | 0.24
Statistical Analysis 1: Comparison: Azacitidine vs Conventional Care; Test type: Superiority or Other; p = 0.1327, exact binomial; Risk Ratio (RR) = 0.67, 95% CI 2-sided [0.35 to 1.20]

14. Secondary Outcome: Number of Participants in Different Categories of Adverse Experiences During Core Study Period
Description: Patient counts for a variety of subsets of adverse experiences for the core study period (day 1 to 42 months). The individual options for Conventional Care Regimens (Best Supportive Care Only, Low-Dose Cytarabine, and Standard Chemotherapy) are presented as separate treatments.
Time Frame: Day 1 (randomization) to 42 months
Population: Safety population excludes 4 Azacitidine patients, 3 Best Supportive Care Only patients, 5 Low-dose Cytarabine patients, and 6 Standard Chemotherapy patients who were randomized/assigned to those regimens but did not receive treatment.
Measure: Number; unit: participants
Groups:
- Azacitidine: Azacitidine, 75 mg/m2/day given by subcutaneous injection for 7 days of every 28 day cycle, plus best supportive care.
- Best Supportive Care Only: Care can include transfusions, antibiotics, myeloid growth factors [G-CSF and GM CSF] for neutropenic infections until the end of the study.
- Low-dose Cytarabine: Cytarabine, 20 mg/m2/day subcutaneously on Days 1-14, with 28-42 days between cycles. Plus best supportive care.
- Standard Chemotherapy: Induction cycle: Cytarabine infusion 100-200 mg/m2/day on days 1-7 + anthracycline on days 1, 2, 3 Consolidation cycle: Cytarabine infusion 100-200 mg/m2/day for 3-7 days + anthracycline on days 1 and 2 There are 28-70 days between cycles - 1 induction cycle and maximum of 2 consolidation cycles; best supportive care follows the final consolidation cycle.
Arm/Group | Azacitidine | Best Supportive Care Only | Low-dose Cytarabine | Standard Chemotherapy
Number analyzed (Participants) | 175 | 102 | 44 | 19
participants
  Patients with >=1 treatment emergent AE (TEAE) | 175 | 97 | 44 | 19
  Patients with >=1 treatment related TEAE | 169 | 1 | 34 | 19
  Patients with >=1 serious TEAE | 114 | 71 | 27 | 14
  Patients with >=1 serious treatment related TEAE | 43 | 0 | 13 | 13
  Patients w TEAE leading to discontinued treatment | 22 | 4 | 6 | 2
  Patients w TEAE leading to dose reduction | 20 | 0 | 2 | 0
  Patients w TEAE leading to dose interruption | 82 | 0 | 12 | 0

15. Post Hoc Outcome: Kaplan-Meier Estimates for Median Time to Transformation to Acute Myeloid Leukemia (AML) Based on the Last Bone Marrow Assessment
Description: A sensitivity analysis of time to transformation to AML during the entire study was performed based on the last bone marrow assessment. Patients were censored based on the last bone marrow assessment.
Time Frame: Day 1 (randomization) to 42 months
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Azacitidine | Conventional Care
Number analyzed (Participants) | 179 | 179
months | 17.80 [13.6 to 23.6] | 11.48 [8.3 to 14.5]
Statistical Analysis 1: Comparison: Azacitidine vs Conventional Care; Test type: Superiority or Other; p < 0.0001, Log Rank — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Azacitidine vs Conventional Care; Test type: Superiority or Other; p < 0.0001, Regression, Cox; Hazard Ratio (HR) = 0.50, 95% CI 2-sided [0.35 to 0.70] — Cox proportional hazards model stratified on the randomization factors of FAB and IPSS with model term of treatment

16. Primary Outcome: Number of Participants Who Died
Description: Count of participants who died during the study
Time Frame: 42 months
Population: Intent to treat population
Measure: Number; unit: participants
Arm/Group | Azacitidine | Conventional Care
Number analyzed (Participants) | 179 | 179
participants | 82 | 113

ADVERSE EVENTS:
Time Frame: Treatment-emergent AEs for the 'core study' from Day 1 to 42 months.
Description: Safety population excludes 4 Azacitidine patients, 3 Best Supportive Care Only patients, 5 Low-dose Cytarabine patients, and 6 Standard Chemotherapy patients who were randomized/assigned to those regimens but did not receive treatment.
Arm/Group | Azacitidine | Best Supportive Care Only | Low-dose Cytarabine | Standard Chemotherapy
Serious Adverse Events (participants affected / at risk) | 114/175 | 71/102 | 27/44 | 14/19
Other Adverse Events (participants affected / at risk) | 175/175 | 86/102 | 44/44 | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azacitidine (N=175) | Best Supportive Care Only (N=102) | Low-dose Cytarabine (N=44) | Standard Chemotherapy (N=19)
Anaemia (Blood and lymphatic system disorders) | 12 | 3 | 2 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 2 | 0 | 0 | 1
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 19 | 3 | 1 | 5
Haemolysis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 5 | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 2 | 2 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 2 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 0 | 1
Cardiac failure (Cardiac disorders) | 3 | 2 | 1 | 0
Cardiac failure acute (Cardiac disorders) | 2 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 2 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 0 | 1 | 0 | 0
Left ventricular failure (Cardiac disorders) | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 2 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 2 | 0 | 0
Vestibular disorder (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0
Angle closure glaucoma (Eye disorders) | 1 | 0 | 0 | 0
Endophthalmitis (Eye disorders) | 1 | 0 | 0 | 0
Eye Haemorrhage (Eye disorders) | 2 | 0 | 0 | 0
Myopia (Eye disorders) | 1 | 0 | 0 | 0
Retinal artery occlusion (Eye disorders) | 1 | 0 | 0 | 0
Retinal Haemorrhage (Eye disorders) | 1 | 0 | 0 | 0
Retinal tear (Eye disorders) | 1 | 0 | 0 | 0
Strabismus (Eye disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Caecitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Food poisoning (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Ileitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Neutropenic colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Subileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Tooth disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 1 | 0
Catheter site inflammation (General disorders) | 0 | 0 | 1 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0
Death (General disorders) | 0 | 2 | 0 | 0
Facial pain (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0
General physical health deterioration (General disorders) | 2 | 0 | 0 | 0
Injection site nodule (General disorders) | 1 | 0 | 0 | 0
Injection site pain (General disorders) | 1 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 1 | 1
Pain (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 10 | 3 | 5 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0
Abdominal wall abscess (Infections and infestations) | 1 | 0 | 0 | 0
Abscess neck (Infections and infestations) | 1 | 0 | 0 | 0
Arthritis infection (Infections and infestations) | 0 | 0 | 1 | 0
Aspergillosis (Infections and infestations) | 0 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 2 | 0 | 0 | 2
Bronchitis (Infections and infestations) | 1 | 0 | 1 | 0
Bronchopneumonia (Infections and infestations) | 3 | 3 | 0 | 0
Candidiasis (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 2 | 2 | 2 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0 | 0
Corynebacterium infection (Infections and infestations) | 1 | 0 | 0 | 0
Disseminated tuberculosis (Infections and infestations) | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1
Ear infection (Infections and infestations) | 1 | 0 | 0 | 0
Enterobacter bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0
Escherichia sepsis (Infections and infestations) | 0 | 2 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Fungal sepsis (Infections and infestations) | 1 | 0 | 1 | 0
Gasteroenteritis (Infections and infestations) | 1 | 1 | 0 | 0
Gasteroenteritis salmonella (Infections and infestations) | 1 | 0 | 0 | 0
Gingival infection (Infections and infestations) | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 1 | 0 | 1
Klebsiella bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Laryngopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 0
Lung infection (Infections and infestations) | 2 | 0 | 0 | 0
Meningitis (Infections and infestations) | 1 | 0 | 0 | 0
Mucormycosis (Infections and infestations) | 1 | 0 | 0 | 0
Neutropenic infection (Infections and infestations) | 1 | 0 | 0 | 0
Neutropenic sepsis (Infections and infestations) | 4 | 1 | 1 | 2
Oral herpes (Infections and infestations) | 1 | 0 | 1 | 0
Parotitis (Infections and infestations) | 1 | 0 | 0 | 0
Perianal abscess (Infections and infestations) | 2 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 20 | 12 | 2 | 3
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia fungal (Infections and infestations) | 1 | 0 | 0 | 2
Pseudomembranous colitis (Infections and infestations) | 0 | 1 | 0 | 0
Pseudomonal sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0 | 0 | 0
Renal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0
Salmonella sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 6 | 3 | 2 | 0
Septic shock (Infections and infestations) | 3 | 1 | 2 | 0
Sialoadenitis (Infections and infestations) | 1 | 0 | 0 | 0
Splenic abscess (Infections and infestations) | 1 | 0 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0 | 0
Subdiaphragmatic abscess (Infections and infestations) | 1 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 0
Tuberculosis (Infections and infestations) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 5 | 0 | 2 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Synovial rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 3 | 0 | 1 | 0
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Haemosiderosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 30 | 35 | 6 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2 | 1 | 0
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Urinary tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 4 | 3 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 1 | 0
Coma (Nervous system disorders) | 1 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
Grand mal convulsion (Nervous system disorders) | 0 | 1 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Intracranial haematoma (Nervous system disorders) | 0 | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 2 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 2 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal colic (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 2 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urethral stenosis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 2 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Aortic aneurysm (Vascular disorders) | 1 | 0 | 0 | 0
Circulatory collapse (Vascular disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Shock (Vascular disorders) | 0 | 1 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 2 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Azacitidine (N=175) | Best Supportive Care Only (N=102) | Low-dose Cytarabine (N=44) | Standard Chemotherapy (N=19)
Anaemia (Blood and lymphatic system disorders) | 84 | 42 | 19 | 11
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 6 | 8 | 0 | 4
Leukopenia (Blood and lymphatic system disorders) | 31 | 2 | 3 | 6
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 0 | 4 | 0
Lymphopenia (Blood and lymphatic system disorders) | 3 | 0 | 0 | 3
Neutropenia (Blood and lymphatic system disorders) | 114 | 29 | 15 | 10
Thrombocytopenia (Blood and lymphatic system disorders) | 118 | 34 | 21 | 13
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 1
Bundle branch block right (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiomegaly (Cardiac disorders) | 0 | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 6 | 0 | 1 | 1
Chalazion (Eye disorders) | 0 | 0 | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 6 | 1 | 0 | 1
Conjunctivitis (Eye disorders) | 2 | 2 | 2 | 1
Ocular hyperaemia (Eye disorders) | 1 | 0 | 0 | 1
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 21 | 7 | 1 | 5
Abdominal pain upper (Gastrointestinal disorders) | 10 | 3 | 0 | 2
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 2 | 0 | 2 | 1
Constipation (Gastrointestinal disorders) | 88 | 8 | 11 | 8
Diarrhoea (Gastrointestinal disorders) | 38 | 18 | 10 | 12
Dry mouth (Gastrointestinal disorders) | 5 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 10 | 2 | 0 | 2
Gastritis (Gastrointestinal disorders) | 3 | 3 | 0 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 0 | 0 | 2
Gingival bleeding (Gastrointestinal disorders) | 10 | 5 | 2 | 2
Gingival pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Gingivitis (Gastrointestinal disorders) | 6 | 4 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 12 | 5 | 2 | 1
Lip haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Mouth ulceration (Gastrointestinal disorders) | 9 | 6 | 0 | 0
Nausea (Gastrointestinal disorders) | 84 | 12 | 16 | 9
Oral discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Oral soft tissue disorder (Gastrointestinal disorders) | 2 | 1 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 4 | 3 | 2 | 1
Stomatitis (Gastrointestinal disorders) | 5 | 1 | 0 | 2
Vomiting (Gastrointestinal disorders) | 47 | 7 | 5 | 6
Asthenia (General disorders) | 27 | 15 | 12 | 2
Catheter site erythema (General disorders) | 0 | 0 | 0 | 1
Catheter site haematoma (General disorders) | 3 | 0 | 0 | 1
Catheter site haemorrhage (General disorders) | 1 | 0 | 0 | 2
Catheter site pain (General disorders) | 2 | 1 | 1 | 1
Chest pain (General disorders) | 9 | 3 | 2 | 4
Chills (General disorders) | 5 | 2 | 4 | 1
Fatigue (General disorders) | 42 | 11 | 10 | 4
Gait disturbance (General disorders) | 0 | 0 | 1 | 1
General physical health deterioration (General disorders) | 3 | 2 | 0 | 1
Generalised oedema (General disorders) | 1 | 0 | 0 | 1
Injection site bruising (General disorders) | 9 | 0 | 0 | 0
Injection site erythema (General disorders) | 75 | 0 | 0 | 0
Injection site haematoma (General disorders) | 11 | 0 | 3 | 0
Injection site induration (General disorders) | 9 | 0 | 0 | 0
Injection site pain (General disorders) | 32 | 0 | 0 | 0
Injection site rash (General disorders) | 10 | 0 | 0 | 0
Injection site reaction (General disorders) | 51 | 0 | 0 | 1
Mucosal inflammation (General disorders) | 2 | 0 | 2 | 4
Oedema (General disorders) | 9 | 5 | 1 | 3
Oedema peripheral (General disorders) | 23 | 13 | 8 | 3
Pain (General disorders) | 7 | 2 | 1 | 5
Pitting oedema (General disorders) | 3 | 0 | 0 | 1
Pyrexia (General disorders) | 46 | 16 | 17 | 11
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Aspergillosis (Infections and infestations) | 0 | 0 | 0 | 2
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 2
Bacteriuria (Infections and infestations) | 0 | 0 | 1 | 1
Bronchitis (Infections and infestations) | 16 | 8 | 3 | 0
Catheter related infection (Infections and infestations) | 1 | 0 | 0 | 2
Catheter site infection (Infections and infestations) | 0 | 0 | 0 | 2
Clostridial infection (Infections and infestations) | 0 | 0 | 0 | 1
Enterobacter infection (Infections and infestations) | 1 | 0 | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Fungal skin infection (Infections and infestations) | 1 | 0 | 0 | 1
Influenza (Infections and infestations) | 10 | 5 | 1 | 0
Klebsiella bacteraemia (Infections and infestations) | 0 | 0 | 1 | 1
Nail infection (Infections and infestations) | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 33 | 13 | 3 | 0
Oral candidiasis (Infections and infestations) | 11 | 5 | 2 | 1
Oral herpes (Infections and infestations) | 17 | 5 | 1 | 3
Pharyngeal candidiasis (Infections and infestations) | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 8 | 2 | 1 | 1
Pneumonia (Infections and infestations) | 2 | 0 | 3 | 1
Pseudomonas infection (Infections and infestations) | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 5 | 3 | 0 | 1
Rhinitis (Infections and infestations) | 10 | 1 | 1 | 1
Sinusitis (Infections and infestations) | 6 | 1 | 0 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 15 | 4 | 0 | 0
Urinary tract infection (Infections and infestations) | 12 | 3 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 14 | 5 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 5 | 0 | 3 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 4 | 0 | 0 | 1
Scratch (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 19 | 5 | 3 | 1
Alanine aminotransferase increased (Investigations) | 5 | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 1 | 1
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0 | 1
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 2
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 14 | 0 | 2 | 4
Anorexia (Metabolism and nutrition disorders) | 25 | 9 | 5 | 5
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 4 | 2 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 11 | 2 | 1 | 8
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 | 8 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 15 | 7 | 4 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 7 | 5 | 3 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 10 | 5 | 3 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 9 | 3 | 1 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 4 | 4 | 4
Dizziness (Nervous system disorders) | 17 | 7 | 2 | 2
Headache (Nervous system disorders) | 25 | 8 | 6 | 6
Lethargy (Nervous system disorders) | 13 | 2 | 0 | 0
Sinus headache (Nervous system disorders) | 2 | 0 | 0 | 1
Syncope (Nervous system disorders) | 4 | 1 | 1 | 2
Anxiety (Psychiatric disorders) | 9 | 1 | 2 | 3
Depression (Psychiatric disorders) | 9 | 3 | 2 | 1
Hallucination (Psychiatric disorders) | 1 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 15 | 3 | 5 | 4
Sleep disorder (Psychiatric disorders) | 6 | 0 | 0 | 3
Chromaturia (Renal and urinary disorders) | 1 | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 10 | 1 | 0 | 2
Haemoglobinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Nephropathy toxic (Renal and urinary disorders) | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 1
Urethral obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Testicular swelling (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Vaginal inflammation (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 34 | 15 | 5 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 26 | 5 | 7 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 9 | 1 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 26 | 14 | 6 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 3
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 11 | 3 | 2 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 7 | 0 | 0 | 3
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 8 | 7 | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 13 | 3 | 1 | 2
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 20 | 4 | 7 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 20 | 2 | 2 | 3
Purpura (Skin and subcutaneous tissue disorders) | 4 | 1 | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 18 | 1 | 1 | 5
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 7 | 3 | 0 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 1
Arteriosclerosis (Vascular disorders) | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 21 | 10 | 6 | 1
Hypertension (Vascular disorders) | 15 | 4 | 6 | 3
Hypotension (Vascular disorders) | 10 | 2 | 0 | 4
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
Pallor (Vascular disorders) | 4 | 1 | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 2 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator shall have the right to publish and/or present study data provided that the investigator shall (i) furnish the sponsor a copy of any proposed publication or presentation generally thirty (30) days in advance of the submission, (ii) delete any confidential information of the sponsor, and (iii) delay submission for generally up to ninety (90) days to permit the preparation and filing of intellectual property applications or until sponsor gives its consent in a timely manner.